CLINICAL TRIAL: NCT04162158
Title: Safety and Efficacy of Allogeneic NK Cells Therapy in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Collaborators: Shenzhen Third People's Hospital (Other); The first People's Hospital of Zhengzhou (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: beijing302-NK-HCC
Record Dates: First submitted 2019-08-06; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted drug combined with allogeneic NK cell treatment group (Experimental): In addition to traditional symptomatic supportive treatment, Sorafenib, regolfinib or levabinib will be administered in combination with allogeneic NK cells (3 cycles).
  Interventions: Biological: allogeneic NK cells therapy
- Targeted drug treatment group (No Intervention): Sorafenib, regolfinib or levabinib will be administered in addition to traditional symptomatic supportive care.

INTERVENTIONS:
Biological: allogeneic NK cells therapy — PBMC was isolated from the peripheral blood of the donors and infused to the patient after 14 days incubation. In each cycle, patients will be infused 4.0-5.0×10'9 allogeneic NK cells. All patients in the experimental group received a total of three cycles of treatment with one month interval between each treatment.
  Arms: Targeted drug combined with allogeneic NK cell treatment group

SUMMARY:
This is a multicenter, open-label, paired control study to evaluate the safety and clinical efficacy of allogeneic NK cells combined with targeted drug in the treatment for advanced HCC.

DETAILED DESCRIPTION:
Since killer cell immunoglobulin-like receptor (KIR) mismatch can inhibit the negative regulatory signal of autologous major histocompatibility complex (MHC) molecules and ensure sufficient NK cell activation, allogeneic NK cells therapy, as a potential therapeutic option for tumor, has achieved good results in patients with acute myeloid leukemia. In this study, investigators evaluate the safety and efficacy of allogeneic NK cells in the treatment of advanced HCC. 200 patients from three hospitals will be enrolled in this study and followed up for 1 year. Peripheral blood mononuclear cells (PBMCs) were isolated from patient-related donor and cultured in vitro for 15 days and infused to the patient in two consecutive days. Clinical data and laboratory data were collected and analyzed, including survival, impact indicators, hematology, biochemical indicators, and immunological indicators to evaluate the safety and efficacy of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* According to the 2010 edition of the diagnostic criteria for primary liver cancer BCLC, the patient was diagnosed as advanced hepatocellular carcinoma by pathology and imaging (BCLC C phase);
* Child-Pugh A/B (5-9), Eastern Cooperative Oncology Group (ECOG) PS score less than 2 points;
* Laboratory criteria:

  1. Liver function: Child A/B, ALT < 200 U/L, AST < 200 U/L, Tbil <51μmol/L
  2. Renal function: Creatinine clearance ≥ 60ml/minute
  3. Hematologic function: PLT ≥40×10'9/L, WBC ≥2×10'9/L, HGB>80 g/L
  4. Cardiac function: No abnormality in cardiac enzyme and ECG
* Survival expectation is greater than 6 months;
* Patients with active hepatitis B or C were treated with the appropriate NA or DAA medication, and all patients enrolled in the group were treated with targeted drugs.
* The patient has a donor who meets the donor enrollment criteria and all patients and donors sign the Informed Consent Form;

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Co-infected with hepatitis A, hepatitis E, AIDS or other infectious diseases.
* Patients with serious complications such as acute infection and gastrointestinal bleeding within 30 days.
* Patients with other serious systemic and psychiatric diseases.
* Exposure to any cell therapy such as, but not limited to CIK, DC, CTL , PD-1 and stem cells therapy 6 months prior to study drug administration.
* Other conditions that researchers believe may increase the risk of subjects or lead to affected study results, such as the presence of mental illness in subjects.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | From the date of enrollment to the end of two years of follow-up.
  Incidence of Treatment-Emergent Adverse Events as assessed by [National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0]
Overall survival | From the date of enrollment to the end of two years of follow-up.
  Overall Survival (OS) defined as the time from randomisation until death by any cause. Participants will be followed up for survival follow up for at least five years.

SECONDARY OUTCOMES:
Disease control rate | From the date of enrollment to the end of two years of follow-up.
  According to the RECIST criteria, patients with complete response (CR), partial response (PR), and stable disease (SD) were imaged.

CONTACTS AND LOCATIONS:
Overall Officials: Fusheng Wang, Study Chair — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China